CLINICAL TRIAL: NCT01429428
Title: Randomized and Controlled Study About Efficacy and Safety of Far-Infra Red Radiation Emitted by Compression Stockings for Cellulitis Treatment
Brief Title: Far-IR Emitted by Compression Stockings for Cellulitis Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Edileia Bagatin, M.D., PhD - Professor, Federal University of São Paulo
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SIGVARIS; SigvarisUnifesp (Other Grant/Funding Number: Sigvaris do Brasil)
Record Dates: First submitted 2011-08-28; First posted 2011-09-07 (Estimated); Last update posted 2011-09-07 (Estimated); Status verified 2011-09

CONDITIONS: Cellulitis; Quality of Life
Keywords: Cellulitis; Skin ultra-sound images; Treatment; Infra-red light
MeSH Terms: conditions — Cellulitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stockings side one (Placebo Comparator): This side of the compression stockings is just the fabric (placebo).
  Interventions: Other: No far-IR compression stockings
- Stocking side two (Active Comparator): This side of compression stocking emits far-IR radiation.
  Interventions: Other: Far-IR compression stockings

INTERVENTIONS:
Other: Far-IR compression stockings — The far-IR side of compression stocking will be used by subjects, during the day, for six hours a day, during 90 days.
  Arms: Stocking side two
Other: No far-IR compression stockings — This side of compression stocking without far-IR radiation will be used by subjects, during the day, for six hours a day, during 90 days.
  Arms: Stockings side one

SUMMARY:
This is a randomized and controlled study to investigate if the far-IR radiation emitted by compression stockings fabric may be effective and safe as adjuvant treatment for cellulitis that affects the majority of women after puberty.

The investigators expect that the far-IR effects on superficial microcirculation,deep dermis and subcutaneous fat may attenuate the clinical aspect of cellulitis.

DETAILED DESCRIPTION:
Cellulitis is a sex-specific, anatomic and normal condition affecting women after puberty.The main clinical aspect is the irregularity on skin surface which is classified in 4 grades, 0 to III, according to Nurenberg classification, 1978.

It is a multifactorial condition, involving: herniation of subcutaneous fat into deep dermis; vertical fibrous septum from fatty tissue to dermis; alterations in microcirculation; hormonal and inflammatory factors Clinical evaluation is very difficult and the best methods are: high resolution ultrasound and magnetic resonance.

There is no effective management. Many devices have been introduced to treat that aesthetic condition which causes a great discomfort to women. There are few controlled studies with high level methodology and consistent conclusions.

The far-IR radiation can be obtained by low energy emitting devices and its main effects are the interaction with water and temperature increase. This method had already shown efficacy for circulation system disorders and wound healing by activation of TGF-beta and fibroblasts.

Our aim is to evaluate the benefits of far-IR for cellulitis control.

ELIGIBILITY:
Inclusion Criteria:

* Signed Consent Form
* Healthy women
* Age: 25 to 40 years
* Presence of cellulitis - II or III
* No treatment for cellulitis in the last 6 months

Exclusion Criteria:

* Pregnancy
* Vascular disease
* Psychiatric disorder

Ages: 25 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2011-07; Primary Completion 2011-11 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
Changes in ultra-sound images | 0, 30, 60 and 90 days
  High resolution ultra-sound (DemaScan, Cortex Technology, Denmark)is used to measure dermis density and thickness and distance between dermis and fatty tissue in the most evident two areas with cellulitis(thighs and buttocks)

SECONDARY OUTCOMES:
Changes in Cellulitis clinical grade | 0, 30, 60 and 90 days
  Main investigator evaluates the clinical aspect of cellulitis, i.e., the level of irregularity of skin surface, according to Nuremberg and Müller classification in four grades:
  0: no alterations I: alterations only visible by pinching the skin or contracting the muscles II: skin orange or padded aspect is visible when the woman stands up or by pinching the skin or contracting the muscles III: the same alterations of II associated to skin elevations and nodulations
Subject evaluation | day 90th
  Study subjects will give their opinion about modification on cellulitis appearance using a 5-point scale: much worse; worse; no change; better; much better
Changes in Anthropometric measures | 0, 30, 60 and 90 days
  The circumference of thighs, hip and waist are measured in standardized points
Changes in Photographies | 0, 30, 60 and 90 days
  By using the OMNIA device standardized photos are taken in three positions: front buttocks and side view of thighs
Changes in Skin viscoelasticity | 0, 30, 60 and 90 days
  Skin elasticity is measured by suction with the Cutometer device(Courage&Khazaka, Germany) in the most evident two areas with cellulitis(thighs and buttocks)
Changes in DLQI scores | 0 and 90 days
  The application of the quality of life generic questionnaire named Dermatology Life Quality Index or DLQI(Finlay, 1994), version DLQI-Brasil (Ferraz, 2006) will be used to evaluate the impact of cellulitis and its treatment on women´s life
Occurence of adverse events | 30, 60 and 90 days
  Report and/or observation of side effects,such as discomfort, difficulty to use the stockings or any distress will be registered
Occurence of venous insufficiency signs | 30, 60 and 90 days
  Symptoms and signals of venous insufficiency such as fatigue, swelling, burning will be evaluate by a five-point scale:0=none; 1 = slight; 2 = slight to moderate; 3 = moderate to severe; 4 = severe; 5 = unbearable
Changes in Colour eco-doppler | 0 and 90 days
  Superficial and deep venous systems will be evaluate before and at the end of the study by colour eco-doppler

CONTACTS AND LOCATIONS:
Overall Officials: Edileia Bagatin, M.D., PhD, Principal Investigator — Universidade Federal de Sao Paulo, Brasil